CLINICAL TRIAL: NCT05905133
Title: A Multi-Center, Single-Arm, Open-Label Clinical Study to Evaluate the Safety and Efficacy of CBP-201 in Chinese Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety and Efficacy of CBP-201 in Chinese Adult Subjects With Moderate to Severe AD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBP-201-CN003
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBP-201 (Experimental): The subjects will receive CBP-201 600 mg (4 mL in total, 2 injections of 2 mL each in different sites) on Day1, begin to receive a subcutaneous injection of CBP-201 300 mg (2 mL) from Week2, and receive CBP-201 300 mg (2 mL) every 2 weeks thereafter until Week10.
  Interventions: Drug: CBP-201

INTERVENTIONS:
Drug: CBP-201 — subcutaneous injection
  Other Names: CBP-201 injection

SUMMARY:
This study is a single-arm, open-label, multi-center clinical study designed to assess the safety and efficacy of CBP-201 in eligible subjects with moderate to severe Atopic Dermatitis.

DETAILED DESCRIPTION:
The study includes a screening period, a treatment period and a follow-up period.

The subjects will receive a subcutaneous injection of CBP-201 600 mg (4 mL in total, 2 injections of 2 mL each in different sites) on Day1, begin to receive a subcutaneous injection of CBP-201 300 mg (2 mL) from Week2, and receive CBP-201 300 mg (2 mL) every 2 weeks thereafter until Week10.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ age ≤ 75 years at the screening visit, male or female.
2. Diagnosed with atopic dermatitis (according to the American Academy of Dermatology's Guidelines of care for the management of atopic dermatitis, 2014[1]) at the time of screening, and meeting all the 4 criteria below:

   1. Suffering from the disease for more than 1 year at the time of screening;
   2. At the screening and baseline visit, IGA score ≥ 3 (according to the validated Investigator Global Assessment for Atopic Dermatitis [vIGA-AD™] scale);
   3. EASI score ≥ 12;
   4. Percentage of total BSA affected by AD ≥ 10%.
3. Female subjects of childbearing potential (FCBP) and male subjects who have not undergone vasectomy must agree to take highly effective contraceptive measures during the entire study period (from the signing of informed consent forms (ICFs) to the 8-week follow-up period after discontinuation of study drug). Postmenopausal women (determined by testing follicle stimulating hormone [FSH]; defined as the women who have had amenorrhea for at least 12 consecutive months without using drugs known to cause amenorrhea, and have a recorded FSH level greater than 40 mIU/mL or in the postmenopausal range) and women with a record of surgical sterilization (i.e., tubal ligation or hysterectomy or bilateral oophorectomy) before the screening visit can be considered infertile.

   Highly effective contraceptive measures include:

   i. Abstinence (acceptable only if it is part of the subject's routine lifestyle); ii. Hormones (oral, patch, ring, injection, implant) combined with male condoms. This measure must be used at least 30 days before the first study drug administration. Otherwise, another acceptable method of contraception must be used; iii. Intrauterine device (IUD) combined with male condoms.
4. Subjects are willing and able to comply with study visits and related procedures.
5. Subjects have the ability to learn the study requirements and process, and voluntarily take part in the clinical trial and sign an ICF.

Exclusion Criteria:

1. Received prior treatment with anti-interleukin-4 receptor α (IL-4Rα)/anti-interleukin-13 (IL-13) antibodies with a poor response (including treatment failure or development of unacceptable treatment-related adverse reactions).
2. Have received any of the following topical treatments within 2 weeks before D1 visit: phosphodiesterase-4 (PDE-4) inhibitors, Janus kinase (JAK) inhibitors, or aromatic hydrocarbon receptor agonists.
3. Have received systemic treatment with corticosteroids (except for corticosteroid inhalers and nasal sprays) or other immunosuppressive/immunomodulatory agents (including but not limited to cyclosporine, mycophenolate mofetil, azathioprine, methotrexate, JAK inhibitors, and various biological agents) within 2 weeks before D1 visit or 5 drug half-lives (if known), whichever is longer.
4. Have received treatment with immune cell depletion agents (e.g., rituximab) within 6 months before D1 visit.
5. Have received any investigational drug/treatment within 4 weeks before D1 visit or 5 drug half-lives (if known), whichever is longer.
6. Other skin complications in addition to AD that may interfere with the study assessments.
7. There is a known or suspected history of immunosuppression/immunodeficiency within 6 months before D1 visit (including but not limited to a history of invasive opportunistic infections, such as aspergillosis, coccidiosis, histoplasmosis, acquired immunodeficiency syndrome (AIDS), listeriosis, or Pneumocystis, even if the infection has subsided), or there is an abnormally frequently recurrent or persistent infection.
8. Received systemic treatment with anti-infective drugs (including but not limited to antibiotics, antiviral drugs, antiparasitic drugs, antiprotozoal drugs, or antifungal drugs) due to acute or chronic infection within 1 week before D1 visit (after the infection subsides, the subjects can be rescreened).
9. History of malignant tumor within 5 years before D1 visit (except for completely cured cervical carcinoma in situ or non-metastatic cutaneous squamous cell carcinoma or basal cell carcinoma).
10. History of parasite infection within 6 months before D1 visit.
11. Positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) and HBV-DNA, or positive for hepatitis C antibody and HCV ribonucleic acid (RNA) polymerase chain reaction, or serologically positive for human immunodeficiency virus (HIV) at the screening visit.
12. Subjects with active tuberculosis, latent tuberculosis, or a history of nontuberculous mycobacterial infection at screening;

    Note:
    * Unless there is a clear medical record proving that the subject has received adequate treatment and is currently able to start receiving biological treatment (based on the medical judgment of the investigator and/or infectious disease specialist);
    * If needed, an interferon gamma release assay may be used to assist diagnosis of suspected tuberculosis.
13. Any of the following laboratory test abnormalities at the screening visit:

    1. Aspartate aminotransferase or alanine aminotransferase > 2 times the upper limit of normal (ULN);
    2. Total bilirubin > 1.5 × ULN;
    3. Serum creatinine > 1.2 × ULN;
    4. White blood cell count < 3.0 × 109/L or ≥ 14 × 109/L; Note: If the subjects have the above laboratory test abnormalities at screening, after being assessed as necessary by the investigator, they are allowed to receive a retest on another day within 28 days of the screening period, and those qualified for the retest are permitted to be enrolled (it is forbidden to conduct drug intervention for those laboratory test abnormalities before retest).
14. History of hypersensitivity to L-histidine, trehalose or Tween (polysorbate) 80, or systemic hypersensitivity reactions to any biological agents (except local injection site reactions).
15. History of alcohol or drug abuse within 2 years before D1 visit.
16. Have been vaccinated with (attenuated) live vaccine within 8 weeks before D1 visit, or planning to be vaccinated during the study period.
17. Planning to undergo major surgical operations during the study period.
18. Pregnant or lactating women, or subjects with pregnancy or lactation plans during the study period.
19. Any other conditions (e.g., those may increase the risks of the subjects, or may affect/interfere with the assessment of the study) that the investigator deems unsuitable for participation in this study, including but not limited to: prior or current physical or mental illness, clinically significant physical examination results, vital signs, or safety laboratory test abnormalities at screening. The specific reasons for subjects excluded due to this criterion will be indicated in the study documents (including medical records and electronic case report form (eCRF)).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From Day 1 study drug first administrated to Week 20
  cases/person-years

SECONDARY OUTCOMES:
Incidence of treatment-related treatment-emergent adverse events (TEAEs) | From Day 1 study drug first administrated to Week 20
  cases/person-years
Incidence of serious adverse events (SAEs) | From Day 1 study drug first administrated to Week 20
  cases/person-years
Incidence of treatment-related serious adverse events (SAEs) | From Day 1 study drug first administrated to Week 20
  cases/person-years
Incidence of adverse events of special interest (AESIs) | From Day 1 study drug first administrated to Week 20
  cases/person-years
Abnormal changes in vital signs | Pre-dose, Day1, Day15, Day29, Day43, Day57, Day71, Day85, Day113, Day141
  Vital signs (VS): including body temperature, respiration rate, blood pressure, and heart rate.
Abnormal changes in physical examination | Pre-dose, Day85, Day141
  Physical examination included are as follows: general appearance, skin, ears/nose/throat, head and neck, cardiovascular system, respiratory system, abdomen, limbs, lymph nodes, musculoskeletal and nervous systems.
Abnormal changes in laboratory tests: Hematology | Pre-dose, Day1, Day15, Day29, Day57, Day85, Day141
  White blood cell count, Hemoglobin, Hematocrit, Red blood cell count, Platelet count, Neutrophil percentage, Lymphocyte percentage, Monocyte percentage, Basophil percentage, Eosinophil percentage, Absolute neutrophil count, Absolute lymphocyte count, Absolute monocyte count, Absolute eosinophil count, Absolute basophil count
Abnormal changes in laboratory tests: Blood biochemistry | Pre-dose, Day1, Day15, Day29, Day57, Day85, Day141
  Sodium, Potassium, Calcium, Chlorine, Serum urea/urea nitrogen, Creatinine, Glucose, Total protein, Albumin, Total bilirubin, Alanine aminotransaminase, Aspartate aminotransferase, γ-glutamyltransferase, Alkaline phosphatase, Lactate dehydrogenase, Creatine phosphokinase, Total cholesterol, Low-density lipoprotein, High-density lipoprotein
Abnormal changes in laboratory tests: Urinalysis | Pre-dose, Day1, Day15, Day29, Day57, Day85, Day141
  Urine bilirubin, Urine red blood cells, Urine white blood cells, Urine glucose, Urine ketone, Urine nitrite, Urine pH, Urine protein, Urine specific gravity, Urobilinogen, Microscopic examination (if necessary)
Abnormal changes in electrocardiogram (ECG) parameters | Pre-dose, Day1, Day141
  ECG variables include ventricular heart rate and PR, QRS, QT, and QTcF intervals.
Proportion of subjects achieving greater than or equal to 75% improvement in Eczema Area and Severity Index (EASI-75) | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  The Eczema Area and Severity Index (EASI) scale quantifies the severity and extent of Atopic Dermatitis, as well as the severity of erythema, infiltration, excoriation, and lichenification of the four anatomical regions-head and neck, trunk, upper extremities, and lower extremities.
Proportion of subjects whose Investigator Global Assessment (IGA) score is 0-1 and decreased by ≥ 2 points from baseline | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  The Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD™) Scale is a 5-point classification scale based on the overall appearance of the skin lesions at a specific time point.
Proportion of subjects achieving greater than or equal to 50% improvement in Eczema Area and Severity Index (EASI-50) | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  The Eczema Area and Severity Index (EASI) scale quantifies the severity and extent of Atopic Dermatitis, as well as the severity of erythema, infiltration, excoriation, and lichenification of the four anatomical regions-head and neck, trunk, upper extremities, and lower extremities.
Proportion of subjects achieving greater than or equal to 90% improvement in Eczema Area and Severity Index (EASI-90) | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  The Eczema Area and Severity Index (EASI) scale quantifies the severity and extent of Atopic Dermatitis, as well as the severity of erythema, infiltration, excoriation, and lichenification of the four anatomical regions-head and neck, trunk, upper extremities, and lower extremities.
Proportion of subjects achieving 100% improvement in Eczema Area and Severity Index (EASI-100) | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  The Eczema Area and Severity Index (EASI) scale quantifies the severity and extent of Atopic Dermatitis, as well as the severity of erythema, infiltration, excoriation, and lichenification of the four anatomical regions-head and neck, trunk, upper extremities, and lower extremities.
Proportion of subjects whose IGA score is decreased by ≥ 2 points from baseline | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  The Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD™) Scale is a 5-point classification scale based on the overall appearance of the skin lesions at a specific time point.
Proportion of subjects with IGA score ≤ 2 (equivalent to reaching a low disease activity state) | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  The Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD™) Scale is a 5-point classification scale based on the overall appearance of the skin lesions at a specific time point.
Proportion of subjects whose weekly average Peak Pruritus Numerical Rating Scale (PP-NRS) is decreased by ≥ 3 points from baseline | Day1, Day15, Day29, Day43, Day57, Day71, Day85, Day113, Day141
  Peak Pruritus Numerical Rating Scale (PP-NRS) is a single self-reported item designed to measure the peak pruritus or the "worst" pruritus in the previous 24 hours.
Proportion of subjects whose weekly average Peak Pruritus Numerical Rating Scale (PP-NRS) is decreased by ≥ 4 points from baseline | Day1, Day15, Day29, Day43, Day57, Day71, Day85, Day113, Day141
  Peak Pruritus Numerical Rating Scale (PP-NRS) is a single self-reported item designed to measure the peak pruritus or the "worst" pruritus in the previous 24 hours.
Change and percentage change in the EASI score from baseline | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  The Eczema Area and Severity Index (EASI) scale quantifies the severity and extent of Atopic Dermatitis, as well as the severity of erythema, infiltration, excoriation, and lichenification of the four anatomical regions-head and neck, trunk, upper extremities, and lower extremities.
Change and percentage change in the weekly average PP-NRS from baseline | Day1, Day15, Day29, Day43, Day57, Day71, Day85, Day113, Day141
  Peak Pruritus Numerical Rating Scale (PP-NRS) is a single self-reported item designed to measure the peak pruritus or the "worst" pruritus in the previous 24 hours.
Change and percentage change in the body surface area (BSA) affected by Atopic Dermatitis from baseline | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  The "Rule of Nines" is used to estimate the maximum percentage of Atopic Dermatitis-affected body surface area (BSA): head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%].
Change and percentage change in the Dermatology Life Quality Index (DLQI) score from baseline | Day1, Day15, Day29, Day57, Day85, Day113, Day141
  Dermatology Life Quality Index (DLQI) is a questionnaire containing 10 items to assess the impact of Atopic Dermatitis on quality of life (QOL) in the past week, and the scores range from 0 (no disease) to 30 (severe disease); the higher the score, the worse the quality of life.
Proportion of subjects receiving concomitant medications for the treatment of the disease under study (Atopic Dermatitis) | from Day1 to Week12
  except emollients; the proportion will be summarized separately by all concomitant medications and the ATC2 codes for concomitant medications
Proportion of subjects receiving concomitant medications for the treatment of the disease under study (Atopic Dermatitis) prohibited by the protocol | from Day1 to Week12
  (except emollients; the proportion will be summarized separately by all concomitant medications, local therapy, systemic treatment, and the ATC2 codes for concomitant medications)
Proportion of subjects receiving topical corticosteroids (TCS) for the treatment of the disease under study (Atopic Dermatitis) | from Day1 to Week12
  If topical corticosteroids (TCS) is considered necessary by the investigator.
Duration of TCS use for the treatment of the disease under study (Atopic Dermatitis) | from Day1 to Week12
  days/person-years
Percentage of subjects positive for anti-drug antibody (ADA) and ADA titer range | Day1, Day15, Day29, Day57, Day85, Day141
  Descriptive statistics will be used to summarize the baseline values of related measurements (ADA, NAb) and the changes from baseline to each visit.
Percentage of subjects positive for neutralizing antibody (NAb) in subjects positive for ADA | Day1, Day15, Day29, Day57, Day85, Day141
  Descriptive statistics will be used to summarize the baseline values of related measurements (ADA, NAb) and the changes from baseline to each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Suzhou Connect, Study Director — Connect Biopharm LLC
Locations (38):
- China (38):
  - Connect Investigative Site 01, Beijing, Beijing Municipality
  - Connect Investigative Site 41, Beijing, Beijing Municipality
  - Connect Investigative Site 14, Fuzhou, Fujian
  - Connect Investigative Site 25, Fuzhou, Fujian
  - Connect Investigative Site 03, Guangzhou, Guangdong
  - Connect Investigative Site 11, Guangzhou, Guangdong
  - Connect Investigative Site 13, Guangzhou, Guangdong
  - Connect Investigative Site 20, Guangzhou, Guangdong
  - Connect Investigative Site 22, Shenzhen, Guangdong
  - Connect Investigative Site 31, Nanning, Guangxi
  - Connect Investigative Site 16, Haikou, Hainan
  - Connect Investigative Site 17, Haikou, Hainan
  - Connect Investigative Site 19, Nanyang, Henan
  - Connect Investigative Site 27, Wuhan, Hubei
  - Connect Investigative Site 28, Yichang, Hubei
  - Connect Investigative Site 26, Changsha, Hunan
  - Connect Investigative Site 34, Nanjing, Jiangsu
  - Connect Investigative Site 39, Suzhou, Jiangsu
  - Connect Investigative Site 05, Zhenjiang, Jiangsu
  - Connect Investigative Site 29, Shenyang, Liaoning
  - Connect Investigative Site 40, Jiangxi, Nanchang
  - Connect Investigative Site 24, Baotou, Nei Monggol
  - Connect Investigative Site 18, Yinchuan, Ningxia
  - Connect Investigative Site 30, Dongying, Shandong
  - Connect Investigative Site 21, Jinan, Shandong
  - Connect Investigative Site 35, Jinan, Shandong
  - Connect Investigative Site 36, Shanghai, Shanghai Municipality
  - Connect Investigative Site 10, Taiyuan, Shanxi
  - Connect Investigative Site 06, Xi’an, Shanxi
  - Connect Investigative Site 15, Yuncheng, Shanxi
  - Connect Investigative Site 23, Chengdu, Sichuan
  - Connect Investigative Site 02, Tianjin, Tianjin Municipality
  - Connect Investigative Site 09, Ürümqi, Xinjiang
  - Connect Investigative Site 07, Hangzhou, Zhejiang
  - Connect Investigative Site 08, Hangzhou, Zhejiang
  - Connect Investigative Site 33, Hangzhou, Zhejiang
  - Connect Investigative Site 37, Hangzhou, Zhejiang
  - Connect Investigative Site 32, Ningbo, Zhejiang